CLINICAL TRIAL: NCT04954001
Title: A Multi-center, Open-label, Single-arm Phase I Dose-escalation and Phase II Dose-expansion Study to Evaluate the Safety, Tolerability, PK Characteristics and Anti-tumor Activity of FCN-159 in Adult and Pediatric Participants With Neurofibromatosis Type 1
Brief Title: Study to Evaluate the Safety, Tolerability, PK Characteristics and Anti-tumor Activity of FCN-159 in Adult and Pediatric Participants With Neurofibromatosis Type 1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-002
Record Dates: First submitted 2021-06-17; First posted 2021-07-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: FCN-159

INTERVENTIONS:
Drug: FCN-159 — FCN-159 is administered orally in once daily schedule for 28 days a cycle.

SUMMARY:
FCN-159 is a highly active MEK1/2 inhibitor that was designed, synthesized and screened on the basis of the structure of trametinib. FCN-159 is an orally available and highly potent selective inhibitor of MEK1/2, which is expected to be a targeted therapy for the treatment of advanced solid tumors and neurofibromatosis type 1.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria for Phase I and II:

1.Cohort 1: 16-70 years of age (inclusive) with a body weight of ≥ 94 lbs or 42.5 kg.

Cohort 2: 2-15 years of age (inclusive) and able to swallow whole tablet. 2.Participants must be diagnosed with NF1-related plexiform neurofibromas (PN) and symptomatic with requirement of systematic therapy per investigator's judgment. A PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal PN involves two or more levels with connection between the levels or extending laterally along the nerve. Diagnosis of neurofibromatosis type 1 (NF1) is based on meeting at least 1 of the following 2 diagnostic criteria:

1. Genetic testing confirmation: i.e., positive for NF1 germline mutation per CLIA-certified laboratory (or equivalent) testing. Note: NF1 germline mutation positive must either be confirmed by the FCN-159-002 central laboratory or have documentation of NF1 mutation issued by a CLIA-certified laboratory (or equivalent) - OR -
2. Clinical and imaging confirmation: Meets at least 2 of the following 7 NF1 diagnostic criteria according to the clinical NIH consensus criteria:

   1. ≥ 6 cafe-au-lait macules (>0.5 cm in prepubertal participants and > 1.5 cm in post-pubertal participants);
   2. Axillary freckling or freckling in inguinal regions;
   3. ≥2 neurofibromas of any type, or ≥ 1 plexiform neurofibroma;
   4. An optic pathway glioma;
   5. ≥2 Lisch nodules (iris hamartomas);
   6. A distinctive bony lesion such as dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex);
   7. First-degree relative with NF1. 3. Participants should meet one of the following criteria

   <!-- -->

   1. Must be judged by the investigator to be inoperable for complete resection without causing substantial damage, or unsuitable for surgery with high surgical risks , e.g. due to encasement of or close proximity to vital structures, invasiveness, or high vascularity、Extensive lesion scope surgery is not feasible. NF1 has to cause or has the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, paraspinal lesions that can cause myelopathy, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or are significantly disfiguring, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions.
   2. The participants who have previously received surgical treatment, if the PN resection is incomplete, the postoperative residual exceeds 15% of the primary lesion, or relapse after surgery, and the lesions of at least 3 cm are measured in one dimension, are eligible for enrollment. At least a 28-day interval is required between surgery and the first dose of FCN-159.

      4. Participants must have a measurable lesion, defined as at least 3 cm in length in at least one dimension, amenable to MRI for efficacy assessment.

      5. Adult participants: Karnofsky performance level of ≥70%; Pediatric participants: Lansky performance score ≥ 70%, see Appendix 18.

      Note: Participants who are wheelchair bound because of paralysis secondary to a plexiform neurofibroma should be considered ambulatory when they are in the wheelchair. Similarly, participants with limited mobility secondary to the need for mechanical support (such as an airway PN requiring tracheostomy or CPAP) will also be considered ambulatory for the purposes of this study.

      6. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN.

      7. Participants or their legal guardians (if the participant is <18 years old) are able to understand and voluntarily sign a written informed consent form.

      8. For participants of childbearing potential: participants must agree to take effective contraception, and receive double barrier contraception, condom, oral or injectable contraceptives, intrauterine device and other contraceptive methods during treatment and for at least 90 days after the last dose. Male participants must agree to avoid sperm donation for at least 90 days after the last dose.

      9. Willing to avoid excessive sun exposure and use adequate amounts of sunscreen if sun exposure is anticipated.

      Exclusion Criteria:

      Participants who meet any of the following conditions shall not be included in this clinical study:

      Exclusion criteria for Phase I and II:
      1. Participants who have previously received one of the following:

         1. Chemotherapy for NF1 within 3 months of enrollment. Ongoing side effects of that treatment > Grade 1 (except alopecia).
         2. Treatment with any drug or biologic therapy within 14 days of starting FCN-159, such as: tipifarnib, pirfenidone, Peg-Interferon, sorafenib or other VEGFR inhibitors
         3. Strong CYP3A4, CYP2C8 and CYP2C9 inhibitors or inducers (moderate inducers for CYP2C8 and CYP2C9) within 14 days before treatment of the study drug, except for topical skin use.
         4. Use of growth factors to increase the number or function of platelets or white blood cells within 7 days before administration of FCN-159.
         5. Radiotherapy, surgery or immunotherapy within 4 weeks before administration of FCN-159.
         6. Participation in other interventional clinical trials within 4 weeks before administration of FCN-159.
         7. Prior treatment with selumetinib or any other MEK 1/2 inhibitors (specific for phase 2 part).
      2. Participants with malignant tumors associated with NF1 requiring chemotherapy, radiotherapy, or surgery, such as intermediate- to high-grade optic gliomas or malignant peripheral nerve sheath tumors.
      3. Patients have other malignant tumor history or with other malignant tumors simultaneously (excluding cured non-melanoma skin basal cell carcinoma, breast carcinoma in situ or cervix cancer in situ, and other malignant tumors without disease evidence for the past 5 years);
      4. Participants who are unable to undergo MRI examination and/or for whom MRI examination is contraindicated (e.g., due to prostheses, orthotics or dental appliances or due to interference with volumetric analysis of target PN on MRI).
      5. Uncontrolled hypertension (despite medical therapy)

         * Adult participants: defined as systolic or diastolic blood pressures > 140/90 mmHg on repeat examination with existing anti-hypertension therapy.
         * Pediatric participants: Blood pressure (BP) greater than or equal to the 95th percentile for age, height, and gender measured as described in (Appendix 19).
      6. Participants with dysphagia, active digestive diseases, malabsorption syndrome, or other conditions that might affect the absorption of the study drug.
      7. Previous or current retinal vein occlusion (RVO), retinal pigment epithelial detachments (RPED), glaucoma and other significant abnormality in ophthalmic examination.
      8. Interstitial pneumonia, including existing clinically significant radiation pneumonitis.
      9. Cardiac dysfunction or concomitant diseases meeting any one of the following conditions will be excluded:

         1. Three 12-lead electrocardiogram (ECG) measurements performed at the study site during the screening period for which the mean value of three measurements was calculated according to the QTcF formula using the instrument, with QTcF > 470 milliseconds; Participants with risk factors for QTcF prolongation, such as uncorrectable hypokalemia, hereditary long QT syndrome; or receiving drugs that prolong QTcF interval (mainly class Ia, Ic, III antiarrhythmic drugs). Drugs with potential to prolong QTcF interval, See Appendix 20.
         2. New York Heart Association (NYHA) Class ≥ 3 congestive heart failure;
         3. Clinically significant arrhythmia, including but not limited to complete left bundle branch block, second degree atrioventricular block;
         4. Known concurrent clinically significant coronary artery disease, cardiomyopathy, severe valvular disease.
         5. Ultrasound Cardiogram performed during the screening showing. Left ventricular ejection fraction LVEF < 50%.
      10. Participants with active bacterial, fungal or viral infections, including active hepatitis B (hepatitis B virus surface antigen positive and hepatitis B virus DNA > 1000 IU/ml or meeting the study site's diagnostic criteria for active hepatitis B infection), hepatitis C (hepatitis C virus RNA positive), or human immunodeficiency virus infection (HIV positive).
      11. Pregnant or lactating women.
      12. Known hypersensitivity to the study drug, other MEK 1/2 inhibitor or its excipients.
      13. Clinically significant condition that, in the opinion of the investigator, would preclude study participation or compliance with safety requirements.
      14. Inability to attend in-person appointments per current clinical site COVID 19 guidelines and restrictions.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety: Dose-limiting toxicity (DLT) incidence rate. | 28 days after the dose of FCN-159 for DLT
Phase I: Safety: MTD and RP2D. | Approximately 6-9 months for MTD and RP2D (phase I duration)
Phase II: Objective response rate (ORR) by investigator assessment | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Phase I Other safety: - The type and frequency of adverse events (AE) - Treatment-Emergent Serious Adverse Events (SAE) - The frequency and causes of death events - Laboratory safety test results - Changes in vital signs | Through study completion, an average of 2 years
Phase I Efficacy: objective response rate (ORR) by investigator /BIRC assessment, clinical benefit rate (CBR) per investigator/BIRC assessment including CR, PR, and SD lasting more than 6 months; | Through study completion, an average of 2 years
Phase I: Maximum Observed Plasma Concentration (Cmax) After Single Dose and Multiple Dose of FCN-159 | Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 10, 24 hours post-dose on Cycle 1 Day 1 (1 cycle = 28 days) for single dose, Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 10, 24 hours post-dose on Cycle 1 Day 28 for multiple dose
Phase I: AUC From Time Zero to Last Measurable Concentration (AUClast) After Single Dose and Multiple Dose of FCN-159 | Pre-dose (0 hour), 0.5~1, 1.5~3, 4~6, 24 hours on Day 1 of Cycles 2, Pre-dose (0 hour) on Cycle 5 and every 4 cycles thereafter (assessed up to 104 weeks) (1 cycle = 28 days)
Phase I PD marker: ERK phosphorylation inhibition in peripheral blood mononuclear cells (PBMCs) | During Cycle 1 (cycle is 28 days): Day 1, Day 8 and Day 28
Phase I Changes in NF1-related symptoms. | Through study completion, an average of 2 years]
  Each participant will undergo standardized functional evaluations according to the relevant category or categories of PN-related complications. The incidence of patients with improved function or quality of life will be measured. Key measurements are chosen from each complication category to assess for change over time.
Phase II: Critical secondary endpoint: Objective response rate (ORR) by BIRC assessment | Through study completion, an average of 2 years
Phase II: Other efficacy endpoints: Clinical Benefit Rate (CBR) | Through study completion, an average of 2 years
  Per investigator/BIRC assessment including CR (Complete Response), PR (Partial Response), and SD (Stable Disease) lasting more than 6 months;
Phase II: Other efficacy endpoints: Disease Control Rate (DCR) | Through study completion, an average of 2 years
  Defined as the percentage of cases with best response (PR or CR or stable disease (SD) after treatment in evaluable cases.
Phase II: Other efficacy endpoints: Progression-Free Survival (PFS) | Through study completion, an average of 2 years
  Defined as the time from participant enrollment to disease progression or death (whichever occurs first). Participants without an event (no progression or death) were censored at the date of last tumor evaluation.
Phase II: Other efficacy endpoints: Time To Progression (TTP) | Through study completion, an average of 2 years
  Defined as the time from participant enrollment to disease progression, and participants without events (without progression or death) were censored at the date of tumor evaluation.
Phase II: Other efficacy endpoints: Time To Response (TTR) | Through study completion, an average of 2 years
  Defined as the time from participant enrollment to the first observation of tumor response among participants with an objective response
Phase II: Other efficacy endpoints: Duration Of Response (DOR) | Through study completion, an average of 2 years
  Defined as the time from first observation of tumor response to tumor progression or death from any cause in participants with an objective response, (whichever occurs first).
Phase II Other safety endpoints: - The type and frequency of adverse events (AE) - Treatment-Emergent Serious Adverse Events (SAE) - The frequency and causes of death events - Laboratory safety test results; - Changes in vital signs; | Through study completion, an average of 2 years
Phase II Dose intensity | Through study completion, an average of 2 years
  Dose intensity, planned dose intensity and relative dose intensity will be measured.
  Dose Intensity (mg/day) = Actual Cumulative Dose (mg)/ Total Duration of Exposure (Days).
  Plan Dose Intensity (mg/day) = Plan Cumulative Dose (mg) / Total Duration of Exposure (Days).
  Relative Dose Intensity (%) = Dose Intensity / Plan Dose Intensity.
Phase II Ctrough After Multiple Dose of FCN-159 | Pre-dose (0 hour), 0.5~1, 1.5~3, 4~6, 24 hours on Day 1 of Cycles 2, Pre-dose (0 hour) on Cycle 5 and every 4 cycles thereafter (assessed up to 104 weeks) (1 cycle = 28 days)
Phase II Clinical outcome variables: Changes in pain intensity. | Through study completion, an average of 2 years
  Each participant will undergo standardized assessments to evaluate changes in pain intensity, using validated pain scales and questionnaires. The incidence of patients experiencing a decrease in pain intensity, as well as the reduction in pain intensity scores, will be evaluated.
Phase II Other clinical outcome variables: Changes in COA variables other than pain intensity. | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Principal Investigator Hans, Gainesville, Florida
  - John Hopkins All Children Hospital, St. Petersburg, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Medical University of South Carolina - Hollings Cancer Center - PPDS, Charleston, South Carolina
- China (6):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Wuhan
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Hu X, Wu Z, Wang J, Li W, Zeng K, Li Y, Tao J, Guan Z, Kang Z, Xu Z, Ma Y, Yang L, Wang X, Han P, Lin H, Diao L, Tan Y, Zhong W, Hui AM, Li C, Lin X. Phase 1 Study of Luvometinib Use in Pediatric Patients with Neurofibromatosis Type 1-Related Unresectable Plexiform Neurofibromas. Target Oncol. 2025 Nov;20(6):991-1001. doi: 10.1007/s11523-025-01176-y. Epub 2025 Oct 26. PMID 41139346
- [Derived] Hu X, Li W, Zeng K, Xu Z, Li C, Kang Z, Li S, Huang X, Han P, Lin H, Hui AM, Tan Y, Diao L, Li B, Wang X, Wu Z, Lin X. Phase 1 dose-escalation study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of FCN-159 in adults with neurofibromatosis type 1-related unresectable plexiform neurofibromas. BMC Med. 2023 Jul 3;21(1):230. doi: 10.1186/s12916-023-02927-2. PMID 37400844